CLINICAL TRIAL: NCT03727646
Title: Pilot Study of Preoperative Nicotinamide Riboside (Vitamin B3) Supplementation in Patients Undergoing Elective Left Ventricular Assist Device (LVAD) Implantation
Brief Title: Nicotinamide Riboside in LVAD Recipients
Acronym: PilotNR-LVAD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Kevin O'Brien, Professor, School of Medicine: Department of Medicine: Cardiology: Clinical, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005431
Record Dates: First submitted 2018-10-16; First posted 2018-11-01 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure，Congestive; Heart Failure New York Heart Association Class IV; Mitochondrial Alteration
MeSH Terms: conditions — Heart Failure | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: This single-center, open-label study will compare blood and myocardial NAD+ levels and other mitochondrial endpoints in participants with end-stage heart failure receiving open-label nicotinamide riboside prior to LVAD implantation to similar endpoints from patients previously undergoing LVAD implantation.
Who Masked: Outcomes Assessor
Masking Description: Study biostatistician will be blinded to group (NR vs. untreated controls)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open-label nicotinamide riboside (Experimental): Participants scheduled to receive an LVAD will be prescribed nicotinamide riboside (NR) according to the following administration schedule:
  Dose Escalation Day 1: 250 mg (1 capsule) twice daily (total daily intake = 500 mg) Day 2: 500 mg (2 capsules) twice daily (total daily intake = 1000 mg) Day 3: 1000 mg (4 capsules) twice daily (total daily intake = 2000 mg)
  Dose Maintenance Day 4: 1000 mg (4 capsules) twice daily Day 5-14 as applicable thru Day Before Surgery: 1000 mg (4 capsules) twice daily
  Washout Day of LVAD Surgery and/or Day 15: None
  Interventions: Dietary Supplement: Nicotinamide riboside
- Baseline controls (No Intervention): Patients previously receiving LVADs, in whom blood and myocardial tissue assays for NAD+ levels and mitochondrial function were performed.

INTERVENTIONS:
Dietary Supplement: Nicotinamide riboside — nicotinamide riboside supplied as 250mg capsules
  Arms: Open-label nicotinamide riboside

SUMMARY:
While preliminary data show that oral nicotinamide riboside (NR) supplementation increases myocardial levels of oxidized nicotine-adenine dinucleotide (NAD+) levels in mice, there has been no direct evidence that suggests oral NR increases NAD+ levels or improves mitochondrial function in human hearts. This Pilot Study is designed to obtain feasibility data for a planned, larger study testing the hypothesis that oral NR supplementation will increase myocardial NAD+ levels and improve cardiomyocyte mitochondrial function in participants with advanced heart failure planned for elective left ventricular assist device (LVAD) implantation. To demonstrate safety and feasibility of NR in this patient population, the investigators propose to enroll 5 participants planned for LVAD implantation in a Pilot Study of NR in which participants will receive NR, up-titrated over 3 days to a final NR dose of 1000mg twice daily. Blood and myocardial tissue analyses collected previously from age- and gender-matched LVAD recipients will serve as controls.

DETAILED DESCRIPTION:
This Pilot Study will examine the following Aims:

Aim 1: Enroll 5 participants scheduled for elective left ventricular assist device (LVAD) placement into an open-label study of nicotinamide riboside (NR).

a. Participants will have labs (including safety panels) drawn at baseline (Day 1), then receive escalating doses of NR to a maximum dose of 1000mg twice daily by Day 3. Participants will be continued on NR at 1000mg twice daily until LVAD implantation surgery.

On the morning of LVAD implantation Surgery (Day 5 or later), participants will have final labs drawn. Samples of fresh cardiac tissue removed from the left ventricular apex during LVAD implantation surgery will be collected in the operating room. The primary analyses will be performed on NR-treated participants who were on the maximum NR dose of 1000mg twice daily for at least 2 days prior to LVAD implantation surgery. The maximum duration of NR administration will be capped at 14 days. If the surgery doesn't happen by then, the participant will be withdrawn from the study.

Aim 2: Determine the effect of NR (as compared to historical controls) on levels of the oxidized and reduced forms of nicotine-adenine dinucleotide (NAD+ and NADH, respectively), mitochondrial function and its regulation through modifications of the epigenome in the failing myocardium.

1. Measure NAD+ and NADH levels in the blood and myocardium of the participants.
2. Assess mitochondrial morphology and function in cardiac tissue using, respectively, electron microscopy (EM) and isolated mitochondria.
3. Determine protein acetylation in the mitochondrial and non-mitochondrial compartments and changes in nuclear gene regulation.

Aim 3: Test the hypothesis that NR improves mitochondrial function and reduces inflammatory response in heart failure (HF) patients receiving NR (as compared to historical controls).

1. Measure mitochondrial function in peripheral blood mononucleated cells (PBMC).
2. Determine the inflammatory response in PBMC.
3. Compare effects on the circulating inflammasome vs. myocardial inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced heart failure.
* Planned elective LVAD implantation surgery with patient agreements for candidacy in place as required by UWMC.
* Hospital inpatient at time of enrollment.
* Ability to undergo Study procedures.
* Willingness/ability to provide informed consent.

Exclusion Criteria:

* Current smoking
* Receiving certain concurrent supplements (to be determined at discretion of the PI). Note that UWMC Nutrition Care standards call for a general multivitamin (1 tab PO daily) as part of the advanced heart failure therapy (AHFT) work-up.
* Known allergies to niacin or nicotinamide.
* Hepatic, renal, endocrine, or neurological disease that disqualify them from consideration for LVAD implantation.
* Inability to perform Study visits or procedures.
* Unwillingness/inability to provide informed consent.
* Women who are currently pregnant or who wish to become pregnant over the course of the study follow-up are not allowed to join this study. This exclusion is built into the LVAD candidate selection process.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O'Brien, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Result] Zhou B, Wang DD, Qiu Y, Airhart S, Liu Y, Stempien-Otero A, O'Brien KD, Tian R. Boosting NAD level suppresses inflammatory activation of PBMCs in heart failure. J Clin Invest. 2020 Nov 2;130(11):6054-6063. doi: 10.1172/JCI138538. PMID 32790648

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Nicotinamide Riboside: Participants scheduled to receive an LVAD will be prescribed nicotinamide riboside (NR) according to the following administration schedule:
  Dose Escalation Day 1: 250 mg (1 capsule) twice daily (total daily intake = 500 mg) Day 2: 500 mg (2 capsules) twice daily (total daily intake = 1000 mg) Day 3: 1000 mg (4 capsules) twice daily (total daily intake = 2000 mg)
  Dose Maintenance Day 4: 1000 mg (4 capsules) twice daily Day 5-14 as applicable thru Day Before Surgery: 1000 mg (4 capsules) twice daily
  Washout Day of LVAD Surgery and/or Day 15: None
  Nicotinamide riboside: nicotinamide riboside supplied as 250mg capsules
Period: Overall Study
Arm/Group | Open-label Nicotinamide Riboside | Baseline Controls
Started | 5 | 0
Completed | 4 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: We did not have the funding to enroll baseline controls.
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-label Nicotinamide Riboside | Baseline Controls | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 5 |  | 5
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Full Range); unit: years] | 35.4 [23 to 65] |  | 35.4 [23 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 5 |  | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 3 |  | 3
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5
LV Ejection Fraction [Mean (Full Range); unit: %] | 20.6 [13 to 27] |  | 20.6 [13 to 27]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participates Experiencing Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: Participants experiencing adverse events during the time they are on the study drug.
  Regarding time frame: Day 1 is the first day that the study subjects start taking the study drug (NR). The participants stop taking the study drug on the day before his/her LVAD surgery (between Days 6 and 14).
Time Frame: from Day 1 receiving NR to the day before LVAD surgery (between Day 6-Day 14)
Population: We did not enroll any baseline control subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Nicotinamide Riboside | Baseline Controls
Number analyzed (Participants) | 4 | 0
Participants | 2 |

2. Primary Outcome: Pre/Post NR Comparison of Maximal Mitochondrial Respiration in PBMCs
Description: Comparison of maximal mitochondrial respiration in PBMCs on the Day of LVAD Surgery Pre- vs Post-NR Administration
Time Frame: from Day 1 receiving NR to the day before LVAD surgery (between Day 6-Day 14)
Population: We did not have the funds to enroll baseline control subjects.
Measure: Mean (Standard Deviation); unit: pmole/min/million cells (O2 consump rate
Arm/Group | Open-label Nicotinamide Riboside | Baseline Controls
Number analyzed (Participants) | 4 | 0
pmole/min/million cells (O2 consump rate
  Pre-NR | 140.8 (31.6) |
  Post-NR | 317.8 (107.6) |

3. Secondary Outcome: Effect of NR on Whole Blood NAD+ Levels
Description: Change in whole blood NAD+ levels from Baseline to Day of Surgery in NR-treated participants
Time Frame: from Day 1 receiving NR to the day before LVAD surgery (between Day 6-Day 14)
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Open-label Nicotinamide Riboside (After Receiving NR): Participants scheduled to receive an LVAD will be prescribed nicotinamide riboside (NR) according to the following administration schedule:
  Dose Escalation Day 1: 250 mg (1 capsule) twice daily (total daily intake = 500 mg) Day 2: 500 mg (2 capsules) twice daily (total daily intake = 1000 mg) Day 3: 1000 mg (4 capsules) twice daily (total daily intake = 2000 mg)
  Dose Maintenance Day 4: 1000 mg (4 capsules) twice daily Day 5-14 as applicable thru Day Before Surgery: 1000 mg (4 capsules) twice daily
  Washout Day of LVAD Surgery and/or Day 15: None
  Nicotinamide riboside: nicotinamide riboside supplied as 250mg capsules
- Baseline (Before Receiving NR): Participants who are enrolled in the study prior to receiving any NR.
Arm/Group | Open-label Nicotinamide Riboside (After Receiving NR) | Baseline (Before Receiving NR)
Number analyzed (Participants) | 4 | 4
ug/mL | 40.625 (11.19266873) | 18.025 (2.662548904)

4. Secondary Outcome: Between-group Comparison of Mitochondrial Respiration (Seahorse Assay) in Isolated Peripheral Blood Mononuclear Cells (PBMCs)
Description: Comparison of mitochondrial respiration (Seahorse assay) in isolated peripheral blood mononuclear cells (PBMCs) on the Day of LVAD Surgery in NR-treated vs. historical control patients
Time Frame: Data collected 6-14 days after study intervention (oral NR) has been initiated.
Population: The control subjects were unfortunately not enrolled so we were unable to make the intergroup comparison.
Measure: Mean (Standard Deviation); unit: pmole/min/million cells (O2 consump rate
Arm/Group | Open-label Nicotinamide Riboside | Baseline Controls
Number analyzed (Participants) | 4 | 0
pmole/min/million cells (O2 consump rate | 317.7895265 (107.6126397) |

5. Secondary Outcome: Between-group Comparison of Whole Blood NAD+ Levels
Description: Comparison of whole blood NAD+ levels on the Day of LVAD Surgery in NR-treated vs. historical control patients
Time Frame: Data collected 6-14 days after study intervention (oral NR) has been initiated.
Population: We unfortunately did not enroll any control subjects, hence were unable to make the intergroup comparison.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Open-label Nicotinamide Riboside | Baseline Controls
Number analyzed (Participants) | 4 | 0
ug/mL | 40.625 (11.19266873) |

ADVERSE EVENTS:
Time Frame: from Day 1 receiving NR to 30 days post-LVAD implantation.
Description: The study patients were on NR for a short period of time and it is extremely difficult to tease out their symptoms of terminal HF versus those from NR administration.
Arm/Group | Open-label Nicotinamide Riboside | Baseline Controls
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/0
Other Adverse Events (participants affected / at risk) | 0/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Nicotinamide Riboside (N=5) | Baseline Controls (N=0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0) — The cardiac arrest was determined by our DSMB to be independent of NR administration.
Death (Nervous system disorders) | 1 (1) | NA — The death resulting from post-LVAD CVA was determined to be unrelated to NR administration by our DSMB.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol: Study Protocol (2018-11-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT03727646/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT03727646/SAP_001.pdf